CLINICAL TRIAL: NCT06121050
Title: Can a Patient in Intensive Care be Visited by His or Her Pet? Feasibility Study.
Brief Title: Can a Patient in Intensive Care be Visited by His or Her Pet?
Acronym: ACCOMPAGNE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 21PH263; 2023-A01439-36 (Other: ANSM)
Record Dates: First submitted 2023-11-02; First posted 2023-11-07 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Intensive Care Patients

STUDY DESIGN:
Intervention Model Description: Patients who can be visited by their pets
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pet visit (Experimental): Intensive care patients visited by their pets for 20 minutes
  Interventions: Other: Pet visit

INTERVENTIONS:
Other: Pet visit — Intensive care patients visited by their pets for 20 minutes

SUMMARY:
Nearly half of all intensive care patients describe symptoms of anxiety and depression after a stay in the ICU, and one in five has genuine post-traumatic stress disorder.

As a result, improving patient experience has become a priority in the ICU, and particular attention is being paid to the need to recreate a familiar environment.

Animal-mediated interventions have been developed for a number of patients over many years. These strategies are widely used with elderly patients, and patients with cognitive or psychiatric disorders, for whom the literature shows benefits on anxiety, mood or objective signs of stress.

In the vast majority of experiments carried out to date, the animals (mainly dogs) were prepared and educated for contact with patients, and their handlers trained in this activity, rather like guide dogs. Visiting a care facility with a patient's own pet is rarely described. It may run up against obstacles related to the animal's behavior or infectious risks, but it is nevertheless authorized in many establishments.

ELIGIBILITY:
Inclusion Criteria:

* Conscious adult patients with a pet (dog/cat).
* Patients with no or no longer hemodynamic or respiratory failure, or undergoing rehabilitation, after resolution of the acute phase or at the end of life.
* Patients affiliated to or entitled under a social security scheme.
* Patient who has given written informed consent to participate in the study.

Exclusion Criteria:

* Non-stabilized acute situation (as assessed by the resuscitator).
* Mechanical or amine ventilation or extrarenal purification.
* Tracheostomy.
* Immunosuppression.
* Carriage of multi-resistant bacteria.
* Behavioral or consciousness disorders.
* Pregnancy.
* Skin wounds, extensive burns exceeding 15% of body surface area, external fixator.
* Guardianship or trusteeship.
* Workload incompatible with the visit
* Patient unable to speak French.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-07-03 (Actual); Primary Completion 2029-03 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Feasibility of visiting the pets | Day 15
  The feasibility of visiting the pets of patients hospitalized in the intensive care unit will be measured by the proportion of patients included in the study for whom at least one visit with their pet was possible. A visit will be considered to have taken place as soon as the patient has had contact with his or her pet.

SECONDARY OUTCOMES:
PANAS | Day 1
  The impact of the animal's visit on the patient's mood will be assessed by variations in the scale Positive and Negative Affect Schedule (PANAS). This self-report scale measures positive (PA) and negative (NA) affect, and is made up of 20 items, 10 of which assess PA and 10 of which assess NA. Each item refers to an adjective, and responses are classified on a 5-point Likert scale, according to how the person felt about the emotion described by the adjective. For each patient, the variation in AP and NA is calculated as follows: (score after visit-score before visit)/score before visit.
Paramedical care | Day 1
  The evaluation of the paramedical care load will be assessed by 2 quantitative indicators:
  * The number of paramedical caregivers mobilized for the reception and care of the pet.
  * The time spent by each member of staff on receiving and caring for the pet, in minutes.
Patient microbiological impact | Day 1
  Search for multi-resistant bacteria on rectal and nasal swabs taken from patients on a routine weekly basis (Meticillin-resistant Staphylococcus Aureus, ESBL-producing Enterobacteria, Vancomycin-resistant Enterococcus, Carbapenemase-producing Enterobacteria).
  Stool analysis, in particular for Clostridium Difficile and Salmonella, and bacterial and parasitic research by multiplex PCR.
Intensive care unity microbiological impact | Day 1
  Surface samples will be taken in conjunction with the operational hygiene team before and after the animal visit, in the room where the visit takes place, in the room of each patient included after discharge, and in the care areas of the intensive care unit. These samples will focus on bacteria, fungi and parasites.
Patient satisfaction | 3 months
  Satisfaction survey

CONTACTS AND LOCATIONS:
Overall Officials: Cindy POKRANDT, Principal Investigator — CHU SAINT-ETIENNE
Locations (2):
- France (2):
  - Centre Hospitalier Ardèche Nord, Annonay
  - Centre Hospitalier de Saint-Etienne, Saint-Etienne

IPD SHARING:
Plan to Share IPD: Undecided